CLINICAL TRIAL: NCT05790148
Title: Precision of Different Scanbodies Used for Direct Digital Impression in Fabrication of Implant Supported Fixed Prosthesis: A Methodologic Clinical Study
Brief Title: Precision of Three Different Scanbodies Used for Direct Digitalization Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kıvanç Akça, Prof. Dr., Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KA-19091
Record Dates: First submitted 2022-12-19; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Prosthesis User; Digitalism
Keywords: digital dentistry; intraoral scanner; implant scanbody

STUDY DESIGN:
Masking Description: Scan post information used for direct digitalization was not shared with the patient during the procedure.
  The investigator, who performed the statistical analysis, did not learn the scan post, in which the primary and secondary data were collected, until all evaluations were completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation precision of different scan-bodies (Other): Three different brand scanbodies (Straumann, Medentika, 3Shape) that applied in same participant group with randomization are used in this clinical study. These three different scan bodies are digitized using an intraoral scanner. Three different temporary restorations are designed in the CAD program and three different bridges are produced with the milling technique using the temporary restoration block. Clinical and analytic evaluations were perform and primarly, seconderly outcomes were achieved.
  Interventions: Device: 3Shape

INTERVENTIONS:
Device: 3Shape — original (Straumann), non-original (Medentika) and generic scan-bodies (3Shape) were utilized for direct digitalization using intraoral scanner with image stitching algorithm. Full contour temporary restorations were fabricated from each digital record, and were evaluated in terms of clinical and analytical.
  Other Names: Straumann (CARES Mono Scanbody; Straumann Holding AG), Medentika (Scanbody 2.generation; MEDENTIKA GmbH, Hügelsheim, Germany) , 3Shape (3Shape A/S, Copenhagen, Denmark)

SUMMARY:
The goal of this clinical trials to evaluate precision of different scanbodies in same participant group. The main guestion it aim to answer is:

1. Are the precision of the three different scanbodies used in direct digitalization the same for the produce of implant-supported prostheses?

Participants are healty and have short edentulous span in posterior region that will receive implant-supported prostheses.

DETAILED DESCRIPTION:
Twenty-five patients receiving two implant supported restorations in treatment of short-span partial edentulism were enrolled into the study. Three different scanbodies, original, non-original and generic, were employed for direct digitalization technique. Full contour PMMA restorations were CAD/CAM fabricated from each digital record, and were evaluated in terms of implant fit, axial- and occlusal-contact. Additionally, patient's impressions for digitalization and delivery procedures were recorded using a visual analog scale. Scanbody scan recordings were subjected to reverse engineering for analytical evaluation of 3D virtual implant positioning.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to voluntarily participate in the study after reading the informed consent form.
* Adult patient over 18 years of age who has completed growth and development
* Partial edentulism in the functional region for a two-implant-supported restoration with two or three occlusal members
* Having a fixed dentition in the opposing arch
* The occlusal relationship between the jaws does not require vertical and horizontal prosthetic treatment.
* Having bone-level implants placed with "straightforward" surgery according to the SAC classification system [248] and without advanced surgical technique

Exclusion Criteria:

* Not voluntarily agreeing to participate in the study after reading the informed consent form
* Having one or more of the conditions for which implant treatment is strictly contraindicated (patients who have received radiation therapy, bone cancer, metabolic disorders)
* Having systemic (steroid therapy, uncontrolled diabetes, immunological disorders, pregnancy) risk factors for implant treatment
* Having local (periodontal discomfort, bruxism, poor oral hygiene) risk factors for implant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Clinical fit | 1 year
  Compatibility between the manufactured restorations and implant
  0: incompatible
  1: compatible
occlusal contact | 1 year
  Restoration occlusal contact with the opposite teeth.
  I.Occlusal Contacts:
  1. Perfect: No need for occlusal contact adjustment,
  2. Acceptable: Minor occlusal contact adjustment is needed,
  3. Correction needed: Major occlusal contact adjustment is needed.
interface contact | 1 year
  Restoration interface contacts with the adjacent teeth.
  II. Interface Contacts:
  1. Perfect: The floss is inserted into the interdental space only under pressure,
  2. Acceptable (1): The contact is slightly tight but the floss is placed under pressure,
  3. Acceptable (2): The contact is slightly weak, the floss is placed in one stroke without applying pressure,
  4. Correction required: Contact is poor and 100 μm metal sheet passes easily.
Analytical measurement of 3D implant positions | 1 year
  Analytical outcomes were obtained from scan bodies using reverse engineering software used to calculate 3D implant positions.

SECONDARY OUTCOMES:
Visual analog scale | 1 year
  Patient impression was done in two clinical stages, registration and restoration delivery, and a scale of five points from 0 to 100 was used. A value of 0 is set to be straightforward and 100 complex. During the registration phase, the patient's anxiety level about the direct digitalization procedure, which was explained in detail before registration, was determined. After the registration, it was asked to evaluate the difficulty of the process. The time spent for adjustment during the restoration delivery phase and the comfort feeling of the restoration after adjustment were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Fatmanur Demir, DDS, Principal Investigator — Hacettepe University Faculty of Dentistry Department of Prosthodontics Ankara, Turkey
Locations (1):
- Hacettepe University Faculty of Dentistry Department of Prosthodontics, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oh KC, Park JM, Moon HS. Effects of Scanning Strategy and Scanner Type on the Accuracy of Intraoral Scans: A New Approach for Assessing the Accuracy of Scanned Data. J Prosthodont. 2020 Jul;29(6):518-523. doi: 10.1111/jopr.13158. Epub 2020 Jun 26. PMID 32133690
- [Result] Passos L, Meiga S, Brigagao V, Street A. Impact of different scanning strategies on the accuracy of two current intraoral scanning systems in complete-arch impressions: an in vitro study. Int J Comput Dent. 2019;22(4):307-319. PMID 31840139

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT05790148/Prot_SAP_000.pdf